CLINICAL TRIAL: NCT05193656
Title: Bladder Cancer Detection Using Convolutional Neural Networks
Acronym: BLAInostic
Status: Recruiting | Type: Observational
Sponsor: Zealand University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SJ-905
Record Dates: First submitted 2021-11-17; First posted 2022-01-18 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Bladder Cancer
Keywords: Machine learning; Artificial intelligence
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Detecting bladder tumor: Patients with hematuria, or previous bladder tumor
  Interventions: Diagnostic Test: Al_bladder

INTERVENTIONS:
Diagnostic Test: Al_bladder — Detection of bladder tumor with help of Artificial intelligence

SUMMARY:
The investigators aim to experiment and implement various deep learning architectures to achieve human-level accuracy in Computer-aided diagnosis (CAD) systems. In particular, the investigators are interested in detecting bladder tumors from CT urography scans and cystoscopies of the bladder in this project.

DETAILED DESCRIPTION:
The investigators aim to experiment and implement various deep learning architectures to achieve human-level accuracy in Computer-aided diagnosis (CAD) systems. In particular, the investigators are interested in detecting bladder tumors from CT urography scans and cystoscopies of the bladder in this project. The investigators want to classify bladder tumors as cancer, non cancer, high grade and low grade, invasive and non-invasive, with high sensitivity and low false positive rate using various convolutional neural networks (CNN). This task can be considered as the first step in building CAD systems for bladder cancer diagnosis. Moreover, by automating this task, the investigator scan significantly reduce the time for the radiologists to create large-scale labeled datasets of CT-urography scans and reduce the false-negative and positive that can happen due to human evaluation cystoscopies.

ELIGIBILITY:
Inclusion Criteria:

* Patients with first time hematuria
* Patients with the control program for previous bladder cancer

Exclusion Criteria:

* Patients with control cystoscope for noncancer suspected disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with micro or macroscopic hematuria
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Comparing standard technique to Machine Learning | 5 years
  The accuracy of Machine learning to detect bladder cancer compared to standard cystoscopy

SECONDARY OUTCOMES:
Detecting accuracy of subtypes of bladder cancer | 5 years
  The abelity of Machine Learning to identify high grad bladder cancer from low grad bladder cancer

CONTACTS AND LOCATIONS:
Overall Officials: Nessn Azawi, phd, Principal Investigator — Zealand University Hospital
Locations (1):
- Zealand University Hospital, Roskilde, Denmark

IPD SHARING:
Plan to Share IPD: No